CLINICAL TRIAL: NCT01177696
Title: VALIDATION OF AN INTERVENTION EFFECTIVE IN GROUPS OF FAMILY CAREGIVERS OF DEPENDENT PATIENTS FOR THEIR APPLICATION IN CENTRES OF PRIMARY HEALTH CARE.
Brief Title: Intervention in Groups of Family Caregivers in Primary Health Care
Acronym: IGFC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Responsible Party: Fundacion para la Investigacion y Formacion en Ciencias de la Salud, Fundacion para la Investigacion y Formacion en Ciencias de la Salud
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRS270A08
Record Dates: First submitted 2010-07-30; First posted 2010-08-09 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Mental Health
Keywords: caregivers; Family Health; Psychotherapeutic; Primary Health Care
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- psychotherapy (Experimental): The study aims to evaluate the effectiveness of an intervention of psychotherapy in improving the mental health of caregivers.
  This intervention is based on theoretical approaches to care adjusted to cognitive theory, in order to be applied in primary health care centres.
  Interventions: Behavioral: Psychotherapeutic intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Psychotherapeutic intervention — A psychotherapeutic intervention will be 8 sessions of 90 minutes in a pilot study groups. This intervention has been initially developed for family caregivers of patients with dementia.
  Other Names: Received usual care.
  Arms: psychotherapy

SUMMARY:
Although Primary Health Care (PHC) Teams are used to deal with prevention and treatment of sanitary problems in adults with chronic diseases, they usually have a lack of experience in development of psychotherapeutic interventions. However, these interventions are the ones that achieve better results to reduce symptomatology and improve emotional state of caregivers.

The study aims to evaluate the effectiveness of an intervention of psychotherapy in improving the mental health and quality of life of caregivers. This intervention is based on theoretical approaches to care adjusted to cognitive theory, in order to be applied in primary health care centres.

To assess a cognitive-behavioural intervention to modify dysfunctional thoughts to properly face the care.

DETAILED DESCRIPTION:
Methods/Design: Design: This is multicentre cross-sectional study, randomized in two parallel groups.

Setting: Two different urban PHC. Study population: 150 caregivers will be included by consecutive sampling. They provide mostly all the assistance to care-dependent familiars receiving attention in PHC Centers. Of chance form 100 caregivers will be assigned to the experimental group and 50 to the group control.

Measurements: Each caregiver will be evaluated on a personal interview. The caregivers' assessment protocol: 1) Assessment of different socio-demographic related to care, and caregiver's personal situation. 2)Care-dependent individuals will also be assessed by Barthel Index and Pfeiffer Questionnaire (SPMSQ). 3)Change in caregivers will be the principal measure: family function (Family APGAR Questionnaire), burden short questionnaire (Short Zarit Burden Interview), quality of life (Ruiz & Baca: 1993 Questionnaire), the Duke-UNK Functional Social Support Questionnaire, the General Health Questionnaire-12, and changes in Dysfunctional Thoughts about caring. 4) Intervention implementation measures will also be assessed.

Intervention: A psychotherapeutic intervention will be 8 sessions of 90 minutes in a pilot study groups. This intervention has been initially developed for family caregivers of patients with dementia.

Discussion: Psychotherapeutic interventions have been proved to obtain better results to reduce symptomatology and improve emotional state of caregivers. Moreover, this intervention has been proved to be effective in a different setting other than PHC, and was developed by professionals of Mental Health. If we found that this intervention is effective in PHC and with our professionals, it would be an important instrument to offer to caregivers of care-dependent patients.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers: They provide mostly all the assistance to care-dependent familiars receiving attention in PHC Centers

Exclusion Criteria:

* Those persons who did not share their place of residence with the relative, or who were impossible to locate either due to a change of address or being admitted to hospital or a nursing home, or on account of the patient's death were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-06 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Change in caregivers will be the principal measure: | Initial and 6 months later
  family function (Family APGAR Questionnaire), burden short questionnaire (Short Zarit Burden Interview), quality of life (Ruiz & Baca: 1993 Questionnaire), the Duke-UNK Functional Social Support Questionnaire, the General Health Questionnaire-12, and changes in Dysfunctional Thoughts about caring.

CONTACTS AND LOCATIONS:
Overall Officials: Rodriguez-Sanchez Emiliano, MD, Principal Investigator — La Alamedilla Health Center, Castilla-León Health Service - SACYL, Salamanca, Spain.; Mora-Simón Sara, Study Chair — La Alamedilla Health Center, Castilla-León Health Service - SACYL, Salamanca, Spain.; Porras-Santos Nieves, Study Chair — La Alamedilla Health Center, Castilla y León Health Service - SACYL, Salamanca, Spain.; Patino-Alonso M. Carmen, MD, Study Chair — Departamento de Estadística. Universidad de Salamanca. Salamanca. Spain.; Recio-Rodríguez José-Ignacio, Study Chair — La Alamedilla Health Center, Castilla-León Health Service - SACYL, Salamanca, Spain; Becerro-Muñoz Concepción, MD, Study Chair — La Alamedilla Health Center, Castilla-León Health Service - SACYL, Salamanca, Spain; Pérez-Arachaederra Diana, Study Chair — La Alamedilla Health Center, Castilla-León Health Service - SACYL, Salamanca, Spain; Gómez-Marcos Manuel-Ángel, md, Study Chair — La Alamedilla Health Center, Castilla-León Health Service - SACYL, Salamanca, Spain; García Ortiz Luís, MD, Study Director — La Alamedilla Health Center, Castilla-León Health Service - SACYL, Salamanca, Spain
Locations (1):
- Primary care Research unit. La Alamedilla health centre, Salamanca, Salamanca., Spain

REFERENCES:
- [Derived] Rodriguez-Sanchez E, Mora-Simon S, Porras-Santos N, Patino-Alonso MC, Recio-Rodriguez JI, Becerro-Munoz C, Perez-Arechaederra D, Gomez-Marcos MA, Garcia-Ortiz L. Effectiveness of an intervention in groups of family caregivers of dependent patients for their application in primary health centers. Study protocol. BMC Public Health. 2010 Sep 17;10:559. doi: 10.1186/1471-2458-10-559. PMID 20849630